CLINICAL TRIAL: NCT02962557
Title: Detecting Post-surgical Respiratory Compromise and Prompting Patients to Self-rescue: An Early Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Ken B. Johnson, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 93779
Record Dates: First submitted 2016-09-06; First posted 2016-11-11 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia
Keywords: ventilatory depression
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): The control group will receive no prompts by the recorded voice.
- Experimental (Experimental): The experimental group will receive playback of recorded verbal prompts to breathe with an optional shoulder shake.
  Interventions: Device: NM3, Phillips Medical, Wallingford CT: verbal prompts to breathe with an optional shoulder shake

INTERVENTIONS:
Device: NM3, Phillips Medical, Wallingford CT: verbal prompts to breathe with an optional shoulder shake — The device used is the NM3 by Phillips Medical, Wallingford CT. The prompting for breaths will include a recorded voice played at 100 decibels played by a speaker placed within 4 feet of the patient's head. If successful breath response is monitored by the patient monitors but no additional subsequent breaths occur within 20 seconds, the verbal prompt will be repeated for the patient to breathe. If the verbal prompting does not result in a breath detected by the patient monitors, the verbal prompt will be repeated within 20 seconds, optionally accompanied by a shoulder shake from the shoulder massager.
  Arms: Experimental

SUMMARY:
This study will explore the feasibility of an idea to use standard, FDA-approved patient monitors to detect ventilatory depression and then play a recorded nurse's voice to prompt patients by name to breathe. The voice prompt will occur in addition to when the traditional alarms are sounded by the monitors. The study device consists of commercially available physiologic monitors, a speaker, and a laptop computer. The physiologic monitors include a pulse oximeter with a motion sensor, capnometer, and nasal airway pressure sensor (built into a nasal cannula). Nasal pressure is a commonly used clinical monitor for sleep apnea detection during polysomnography testing in sleep labs.

DETAILED DESCRIPTION:
This study will explore the feasibility of an idea to use standard, FDA-approved patient monitors to detect ventilatory depression and then play a recorded nurse's voice to prompt patients by name to breathe. The voice prompt will occur in addition to when the traditional alarms are sounded by the monitors. The study device consists of commercially available physiologic monitors, a speaker, and a laptop computer. The physiologic monitors include a pulse oximeter with a motion sensor, capnometer, and nasal airway pressure sensor (built into a nasal cannula). Nasal pressure is a commonly used clinical monitor for sleep apnea detection during polysomnography testing in sleep labs.

The study will be conducted in patients that are admitted to the hospital following surgery. Patients will be monitored during the first 24 hours after surgery, first in the recovery room (post anesthesia care unit, or PACU) and then on the hospital floor. The study will enroll patients with a high likelihood of experiencing ventilatory depression and/or partial to complete airway obstruction. This patient group includes those with known or suspected obstructive sleep apnea and those with surgeries associated with moderate to severe postoperative pain that require significant opioid administration after surgery. The study will compare effectiveness of prompting patients to breathe to that of routine clinical practice in the PACU and hospital floor. The hypothesis is that when compared to standard monitoring and interventions by clinical staff, the digitized breath prompting will prompt patients to breathe more quickly, which will lead to higher oxygen-hemoglobin saturations and respiratory rates throughout the first 24 hours of a patient's hospital stay following surgery.

For patient safety purposes, the experimental design of this study will implement this device as a shadow monitor. Patients will be instrumented with standard physiologic monitors per routine practice in each hospital location (PACU and floor). There will be no change in how clinical staff interacts with patients (i.e. prompting to breathe, checking vital signs, administering medications, assessing patient well-being, etc.) Clinical staff may disable the device at any time if patient comfort or safety are in question.

This study involves use of already cleared medical devices in which they are used in accordance with the indications in the cleared labeling. What is unique is that output from these monitoring devices will be used to prompt a patient directly by name to breathe. The goal of this study is to test the feasibility of the idea that patients will respond to prompts to breathe by a digitized prompting system. If the concept is successful in patients after surgery, as it was for healthy volunteers in previous testing, future research steps would include designing a device and testing it in a clinical trial on patients on the general floor.

ELIGIBILITY:
Inclusion Criteria:

Patients that meet the following criteria will be invited to participate in this study:

1. Patients who undergo surgical procedures associated with a post operative hospital stay of at least 24 hours.
2. Patients with known or suspected obstructive sleep apnea (OSA). Known OSA will be defined as a sleep hypopnea study within the last 10 years that is consistent with OSA. Suspected OSA will be defined as a patient with a screening questionnaire (STOP-Bang) score of 5-8 (A score consistent with a high risk of OSA). The STOP-Bang questionnaire is a built in component of the anesthesia preopreative evaluation in EPIC.

   OR
3. Patients who will undergo surgical procedures associated with significant post operative pain and require opioid analgesics to manage pain. Sample procedures include major extremity surgery, spine surgery, abdominal surgery, and chest surgery that require a post operative in patient hospital stay.

Nurses who meet the following criteria will be invited to participate in this study:

PACU nurses who are in charge of caring for consented patients.

Exclusion Criteria:

1. Patients who are discharged home on the day of surgery.
2. Vulnerable populations including pregnant women, prisoners, and people requiring legally authorized representative for consent
3. There are no exclusion criteria for PACU Nurses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation measured by pulse oximetry (SpO2) | Average and median SpO2 will be measured every 10 minutes for approximately the first 24 hours after surgery during the patient's stay
Breath promoting success rate | Change in respiratory rate from baseline to the period 10 seconds after the breath prompt every 10 minutes for approximately the first 24 hours after surgery during the patient's stay

SECONDARY OUTCOMES:
respiratory rate | Average and median respiratory rate will be measured every 10 minutes for approximately the first 24 hours after surgery during the patient's stay
End-tidal CO2 (etCO2) | Average and median etCO2 will be measured every 10 minutes for approximately the first 24 hours after surgery during the patient's stay

CONTACTS AND LOCATIONS:
Overall Officials: Ken B Johnson, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No